CLINICAL TRIAL: NCT07123584
Title: A Randomized Controlled Trial to Evaluate the Safety and Efficacy of an Oral Supplement in Supporting Vision and Eye Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bio Nature Health (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20686
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Dry Eye; Eye Fatigue
Keywords: Blurred Vision; Red or itchy eyes
MeSH Terms: conditions — Dry Eye Syndromes; Asthenopia; Erythema

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye Empower supplement (Experimental)
  Interventions: Dietary Supplement: Eye Empower
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Eye Empower — A multi-ingredient oral supplement formulated to support eye health. Daily dose (3 capsules).
  Arms: Eye Empower supplement
Dietary Supplement: Placebo — Identical gelatin capsules filled with inert rice flour, administered in the same dosage (3 capsules daily).
  Arms: Placebo

SUMMARY:
This is a 4-week virtual randomized, triple-blinded, placebo-controlled clinical trial evaluating the safety and efficacy of Eye Empower, an oral supplement, in adults aged 45 or older experiencing dry eyes, irritation, and fatigue. Participants take 3 capsules daily and complete self-reported eye health questionnaires weekly.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are male or female
* Age 45 or over
* Self-reported concerns about all three of the following symptoms over the last 4 weeks:

Dry eyes, Irritated eyes, Eye fatigue

- Self-reported concerns about any of the following symptoms over the last 4 weeks: Sensitivity to blue light, Blurred vision, far or near, Red or itchy eyes, Eye inflammation

* Generally healthy - do not live with any uncontrolled chronic diseases
* Willing to avoid using any new prescriptions, over-the-counter medications, supplements, and herbal remedies for the study that target eye health. This includes the use of new prescription eyeglasses or sunglasses
* If taking oral over-the-counter supplements or herbal remedies targeted at eye health, has been consistently taking these for at least 3 months prior to starting the study, and is willing to maintain this routine for the study duration
* Willing to maintain their current diet, sleep schedule, and activity level for the duration of the study.

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including cancer, liver, and mental health-related disorders
* Anyone with diagnosed diabetes (Type I or Type II)
* Planning to undergo any procedure related to their eye health during the study
* Planning to undergo any surgeries or invasive treatments for the study duration
* Has undergone any surgeries or invasive treatments in the last six months
* History of any major illness in the last three months
* Anyone currently taking or has taken a supplement with one or more of the active ingredients in the test product in the last month (e.g., turmeric)
* Started any new medications or supplements that target eye health in the past 3 months
* Anyone with known severe allergic reactions that may require the use of an EpiPen, including but not limited to a shellfish or a latex allergy
* Women who are pregnant, breastfeeding, or trying to conceive currently and for the duration of the study
* Anyone on a medication or herbal supplement that can impact the blood (e.g., blood thinner, anticoagulant, etc.) including but not limited to:

Coumadin (Warfarin) Aspirin Plavix (Clopidogrel)

* Anyone who does not consume animal products for religious and/or personal reasons
* Unwilling to follow the study protocol
* Anyone who has undergone any surgeries or invasive treatments in the last three months or has any planned during the study period
* Anyone with a history of substance abuse
* Anyone who uses illicit drugs, including cannabis
* Anyone who drinks heavily (i.e., 8 or more alcoholic drinks per week for women or 15 or more alcoholic drinks per week for men)

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-06 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change in Eye Health Symptoms (Dryness, Irritation, Fatigue, and Visual Acuity) | Baseline, Week 1, Week 2, Week 3, Week 4
  Assessment of changes in eye dryness, irritation, fatigue, and visual acuity using a self-reported questionnaire administered weekly.

SECONDARY OUTCOMES:
Change in Perceived Overall Eye Health | Baseline, Week 1, Week 2, Week 3, Week 4
  Evaluation of participants' self-reported overall eye health using a standardized questionnaire administered weekly throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States